CLINICAL TRIAL: NCT00916214
Title: Improving Compliance Among Elderly Polypharmacy Users Through Community Pharmacy Based Pharmaceutical Care Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ringkobing Love Apotek (Other)
Collaborators: Ministry of Health and Prevention (Unknown)
Responsible Party: Muhammad Saeed, Ringkøbing Løve Apotek
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RLA Trial
Record Dates: First submitted 2009-06-01; First posted 2009-06-09 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2009-09

CONDITIONS: Polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Pharmaceutical care program

INTERVENTIONS:
Other: Pharmaceutical care program — The pharmaceutical care program consists of 2 elements, that includes individualized medication education and regular follow up

SUMMARY:
The aim of the project is to evaluate effectiveness of a multidimensional pharmaceutical care plan in improving compliance among elderly polypharmacy users at community pharmacy settings. The specific objective of the project is to determine effects of pharmaceutical care program on medication adherence and persistence among elderly polypharmacy users.

ELIGIBILITY:
Inclusion Criteria:

* Both men and woman aged more than 65 years and taking more than 2 drugs

Exclusion Criteria:

* Inhabitants of nursing homes
* People receiving unit dose dispensing of medicine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
change in medication adherence from run-in to the end of phase 1 | 6 months
persistence of mean medication adherence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saeed, Principal Investigator — Ringkøbing apotek
Locations (1):
- Ringkøbing Løve Apotek, Ringkøbing, Denmark